CLINICAL TRIAL: NCT05943626
Title: Timing of Circadian Synchronizers: the TOCS Study
Brief Title: Circadian Intervention to Improve Cardiometabolic Health
Acronym: TOCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Depner, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-60
Record Dates: First submitted 2023-06-12; First posted 2023-07-13 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cardiometabolic Syndrome; Type 2 Diabetes; Sleep; Time Restricted Feeding; Lifestyle Factors; Overweight and Obesity; Insulin Sensitivity; Eating Habit; Sleep Hygiene
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Intermittent Fasting; Overweight; Obesity; Insulin Resistance; Feeding Behavior; Sleep Hygiene

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Group allocation will be blinded to research staff and participants until the conclusion of the baseline segment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Provided with general health information on diet and physical activity.
- Intervention Group (Experimental): Circadian-based intervention focused on timing of light exposure and food intake.
  Interventions: Behavioral: Circadian Intervention

INTERVENTIONS:
Behavioral: Circadian Intervention — The circadian intervention group will receive counseling and instruction to reduce evening and nighttime light exposure, increase morning room light and sunlight exposure, and to finish all food consumption at least 4 hours before bedtime.
  Arms: Intervention Group

SUMMARY:
The overall goal is to examine the efficacy of a circadian intervention in people with overweight and obesity and habitual short sleep duration (HSSD). Participants will undergo a randomized controlled trial, with circadian intervention and control (healthy lifestyle) groups. The circadian intervention is designed to reduce nighttime light exposure and after-dinner snack food intake. Alternatively, the control group will receive basic health information (e.g., physical activity, goal setting, and nutrition when eating out).

DETAILED DESCRIPTION:
The study is a randomized controlled trial with control and circadian intervention groups. Group allocation will be blinded to research staff and participants until the conclusion of the baseline segment. The circadian intervention group will receive counseling and instruction to reduce evening and nighttime light exposure, increase morning room light and sunlight exposure, and complete all food consumption at least 4 hours before bedtime. Participants randomized to control will maintain their habitual food intake and sleep habits in their home environment for ~8 weeks. Both groups will have equal contact time with the study team.

Prior to enrollment participants will complete an clinical overnight sleep disorders screening. Baseline consists of an ~1-week ambulatory real-world monitoring segment. Following baseline participants will be randomized to the control or intervention groups for the 8 week experimental segment. Throughout the study sleep duration will be monitored using an actiwatch wrist-device and a daily electronic sleep log. At the end of the baseline and experimental segments participants will complete overnight laboratory visits to assess insulin sensitivity and circadian timing by oral glucose tolerance test and dim light melatonin onset, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-45 years old; equal numbers of men and women
2. Body mass index (BMI): 25.0-34.9 kg/m2,
3. Sleep Habits: habitual self-reported average total sleep time (TST) <6.5 hours per night for prior 6 months

Exclusion Criteria:

1. Clinically diagnosed sleep disorder or major psychiatric illness
2. Evidence of significant organ dysfunction or disease (e.g., diagnosed diabetes, cardiovascular disease, or kidney disease)
3. Use of prescription drugs or substances known to influence sleep or glucose metabolism
4. Shift-work: current or history of within last year
5. Weight change: >10% of body weight over prior six months
6. Experiencing menopause or post-menopausal
7. Current enrollment in weight loss or physical activity program like the Diabetes Prevention Program
8. Currently pregnant or planning to become pregnant, or currently lactating.
9. Currently smoking
10. Alcohol intake >3 drinks per day or >14 drinks per week

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity change from baseline | Change from baseline to end of the ~8 week experimental segment
  Oral Glucose Tolerance Test (OGTT), Matsuda Index

SECONDARY OUTCOMES:
Timing of central circadian clock change from baseline | Change from baseline to end of the ~8 week experimental segment
  Quantified as dim-light melatonin onset from salivary melatonin samples
Plasma ceramides change from baseline | Change from baseline to end of the ~8 week experimental segment
  Fasting plasma samples will be analyzed for plasma ceramides using targeted metabolomics
Average (per week) nightly total sleep time change from baseline | Analyzed as change from baseline for each week of the ~8 week experimental segment
  Analyzed by wrist-actigraphy
Average (per week) sleep satisfaction change from baseline | Analyzed as change from baseline for each week of the ~8 week experimental segment
  5 point likert scale on daily sleep log (1 = very good; 5 = very poor)
Average (per week) self-reported sleep duration change from baseline | Analyzed as change from baseline for each week of the ~8 week experimental segment
  Daily electronic sleep logs will be used to track sleep and waketimes during the ambulatory monitoring phases of the study
Average (per week) timing of food intake change from baseline | Change from baseline to week 8 of the ~8 week experimental segment
  Time of day 50% of calories are consumed collected by picture based food diaries. Average per week will consist of 2 weekdays and 1 weekend day for baseline and final week of intervention
Average (per week) daytime alertness change from baseline | Analyzed as change from baseline for each week of the ~8 week experimental segment
  5 point likert scale on daily sleep log (1= most alert; 5 = not alert at all)

CONTACTS AND LOCATIONS:
Locations (1):
- College of Health Research Complex--University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No